CLINICAL TRIAL: NCT02395926
Title: To Evaluate Safety and the Pharmacokinetic Characteristics After Oral Administration of HT-003 Compared With Choline Alfoscerate Capsule in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HT-003-01
Record Dates: First submitted 2015-02-10; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-02

CONDITIONS: Healthy Male

ARMS (3):
- R (Active Comparator): Gliatilin soft capsule 400mg, administration 3 times per 1day 8:00 a.m., 14:00, 20:00
  Interventions: Drug: Gliatilin 400mg
- T1 (Experimental): HT-003 600mg, administration 2 times per 1 day 8:00 a.m., 20:00
  Interventions: Drug: Choline CR 600mg
- T2 (Experimental): HT-003 600mg*2tab, administration 1 times per 1 day 8:00 a.m.
  Interventions: Drug: Choline CR 600mg

INTERVENTIONS:
Drug: Choline CR 600mg — HT-003 600mg, administration 2 times per 1 day 8:00 a.m., 20:00
  Arms: T1
Drug: Gliatilin 400mg — Gliatilin soft capsule 400mg, administration 3 times per 1day 8:00 a.m., 14:00, 20:00
  Arms: R
Drug: Choline CR 600mg — HT-003 600mg*2tab, administration 1 times per 1 day 8:00 a.m.
  Arms: T2

SUMMARY:
Choline alfoscerate(L-alfa glycerylphosphorylcholine) is a natural compound found in the brain and breast. Choline alfoscerate contains 40.8% of choline and has a produrig structure and separated by a precursor of choline and nerve cell membrane precursor of acetylcholine glycerophosphate. Choline alfoscerate Colin normalization of nerve pathways, nerve cell membrane play and acetylcholine receptor function secondary symptoms caused by cerebrovascular deficiency and indirectly through activation of metabolism, has a degenerative effect on the brain organic mental syndrome.

Currently marketed oral choline alfoscerate received a geriatric cognitive impairment, secondary symptoms and degeneration, or soft capsule is authorized to prescription drugs for degenerative brain organic mental syndrome caused by cerebrovascular deficiency. Gliatilin soft capsules containing 400 mg per 1 capsule 2-3 times one days're supposed to take when considering optimal convenience and efficiency of the drug in patients with the development of sustained release formulations that can be maintained for a long period of time, a certain concentration is required. Accordingly, the modern drug by reducing the frequency of administration a day circuit is to develop a sustained release formulation of choline alfoscerate HT-003 600 mg medication compliance for the purpose of raising. 2 tablets at a time (600 mg x 2) can be taken one day to 1200 mg is required by taking.

Therefore, for the development of sustained release formulation, the test in healthy adult male volunteers targets choline alfoscerate soft capsule formulation of 400mg 3 times per 1 day and sustained-release tablet 600mg 2time per 1 day, pharmacokinetic properties and safety of a single dose should be evaluated when compared.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects between the ages of 20 and 55 years, inclusive
2. BMI>=19kg/m2, <=27kg/m2

   *body mass index (kg/m2) = weight (kg)/ [(height (m)2)
3. Voluntary written consent by the parties that the ability and willingness to participate during the entire period of the test

Exclusion Criteria:

1. Subjects who has history or clinically significant disease about liver, kidney, digestive, respiratory, musculoskeletal, endocrine, neuropsychiatric, blood•tumor type, cardiovascular disease.
2. A GFR of less than 60ml/min person, calculated by the MDRD (Modification of Diet in Renal Disease)

   ※ MDRD equation (mL/min/1.73m2) : GFR = 175 x Scr-1.154 x age-0.203
3. Systolic blood pressure less than 90 mmHg in vital signs is 150 mmHg or diastolic blood pressure less than 50 mmHg or higher or numerical characters shown equal to at least 100 mmHg
4. Subjects with known for hypersensitivity reaction to components of the investigational drug
5. Subjects who has history of drug abuse, shows positive in urine drug screening test
6. Use of any prescription medication within 14 days prior to study medication dosing or use of any medication such as over-the-counter medication including oriental medication within 7 days prior to study medication dosing
7. Participation in any clinical investigation within 60days prior to study medication dosing
8. Subjects with whole blood donation within 60days, component blood donation within 30days
9. Caffeine-containing beverages (coffee, tea, cola) intake or grapefruit / orange juice who exceed the average daily intake of 4 cups.
10. Subjects who intake average alcohol consumption per week exceeds 140g or cannot be a non-alcohol during the hospital stay.
11. Subjects who exceed the average daily smoke of 10 cigarettes or cannot be a non-smoking during the hospital stay
12. Subjects who cannot limit the choline-containing food (liver, cocoa, bean, chocolate, otmil etc), from admitted to the hospital the day before
13. Subjects who shows positive in serum test (hepatitis B, C, HIV)
14. Subjects with decision of nonparticipation through investigator's review due to laboratory test results or other excuse such as non-responding to request or instruction by investigator

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Cmax | in 24hr after administration
AUClast | in 24hr after administration

SECONDARY OUTCOMES:
baseline-corrected Cmax | in 24hr after administration and before administration
baseline-corrected AUClast | in 24hr after administration and before administration
Tmax | in 24hr after administration and before administration

CONTACTS AND LOCATIONS:
Overall Officials: Jungryul Kim, Ph.D, Principal Investigator — Samsung seoul hospital